CLINICAL TRIAL: NCT04613076
Title: A Collaborative, Computer-assisted, Psycho-educational Intervention for Depressed Patients With Chronic Disease at Primary Care
Brief Title: Technology-assisted Collaborative Care Program for Depressed Patients With Chronic Disease at Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Principal Investigator, Graciela Rojas Castillo, Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1180224
Record Dates: First submitted 2020-10-21; First posted 2020-11-03 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Depression
Keywords: Cluster Randomized Controlled Trial; Depression; Hypertension; Diabetes; Primary Care; Psychotherapy; Cognitive-Behavioral
MeSH Terms: conditions — Depression; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Me cuido y me siento mejor" (Experimental): Patients in the primary care clinics assigned to the intervention will receive eight sessions of a computer-assisted, psycho-educational intervention delivered by trained therapists; structured telephone calls by social worker to monitor clinical progress and treatment adherence; usual medical care for chronic diseases; and access to the project's website, which will be populated with information about the project's aims, the research team, and contact data, along with educational material related to depression, diabetes and hypertension, and healthy lifestyles. Study therapists will receive biweekly and monthly supervision by psychologist and psychiatrist, respectively. A monthly meeting will be held between the PCC team and a member of the research team to ensure continuity of care.
  Interventions: Behavioral: "Me cuido y me siento mejor"
- Enhanced Usual Treatment (Active Comparator): The patients in the primary care clinics assigned to the comparator will receive the usual treatment for depression and their physical conditions -all the guaranteed interventions for people with depression, hypertension, and/or diabetes in primary care, according to the Clinical Guidelines for the Treatment of Depression- and their associated basket of health benefits included in the Regime of Explicit Health Care Guarantees. They will have access to the project's website, which will be populated with information about the project's aims, the research team, and contact data, along with educational material related to depression, diabetes and hypertension, and healthy lifestyles.
  Interventions: Behavioral: Enhanced Usual Treatment

INTERVENTIONS:
Behavioral: "Me cuido y me siento mejor" — A multicomponent, collaborative, computer-assisted, psycho-educational intervention for the management of depressive symptoms in primary care patients with diabetes and/or hypertension.
  Arms: "Me cuido y me siento mejor"
Behavioral: Enhanced Usual Treatment — Enhanced Usual Treatment
  Arms: Enhanced Usual Treatment

SUMMARY:
Background: depression and chronic diseases are frequently comorbid public health problems. However, clinical guidelines often fail to consider comorbidities. This study protocol describes a cluster randomized trial (CRT) aimed to compare the effectiveness of a collaborative, computer-assisted, psycho-educational intervention versus enhanced usual care (EUC) in the treatment of depressed patients with hypertension and/or diabetes in primary care clinics (PCC) in Santiago, Chile.

Methods: two-arm, single-blind, CRT carried out at two municipalities in Santiago, Chile. Eight PCC will be randomly assigned (1:1 ratio within each municipality, 4 PCC in each municipality) to the INTERVENTION or EUC. A total of 360 depressed patients, aged at least 18 years, with Patient Health Questionnaire-9 Item [PHQ-9] scores ≥ 15, and enrolled in the Cardiovascular Health Program at the participating PCC. Patients with alcohol/substance abuse; current treatment for depression, bipolar disorder, or psychosis; illiteracy; severe impairment; and resident in long-term care facilities, will be excluded. Patients in both arms will be invited to use the Web page of the project, which includes basic health education information. Patients in the INTERVENTION will receive eight sessions of a computer-assisted, psycho-educational intervention delivered by trained therapists, a structured telephone calls to monitor progress, and usual medical care for chronic diseases. Therapists will receive biweekly and monthly supervision by psychologist and psychiatrist, respectively. A monthly meeting will be held between the PCC team and a member of the research team to ensure continuity of care. Patients in EUC will receive depression treatment according to clinical guidelines and usual medical care for chronic diseases. Outcome assessments will be conducted at three, six, and twelve months after enrollment. The primary outcome will be depression improvement at six months, defined as ≥ 50% reduction in baseline PHQ-9 scores. Intention-to-treat analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Enrolled in the Cardiovascular Health Program (i.e. currently receiving treatment for diabetes and/or hypertension) at the study primary care clinics.
* Patient Health Questionnaire-9 Item (PHQ-9) score ≥ 15.
* Signed informed consent.

Exclusion Criteria:

* Functional illiteracy (i.e., patients unable to read and comprehend written information, such as the study questionnaires or written informed consent).
* Significant visual and/or auditive impairments (i.e., such as those imposing a serious difficulty to respond the study questionnaires or written informed consent).
* Pregnancy or breastfeeding.
* Cognitive impairment - ineligible patients would give a negative answer to questions "What year is it?" and "Where are we (place/address)?".
* In treatment for bipolar and/or psychotic disorder.
* Current psychological treatment for depression.
* High risk of developing alcohol/substance abuse problems, according to an Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) score ≥ 27.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Depression change | Even though the primary outcome is taken at six-month follow-up, this measure will also be reported at three- and twelve-month follow-up.
  Defined as a 50% reduction in a participant's Patient Health Questionnaire-9 Item (PHQ-9) score compared to the baseline.
  The PHQ-9 minimum and maximum values are 0 and 27 points. Higher scores mean worse outcomes.

SECONDARY OUTCOMES:
Proportion of patients who change their depressive status | Three-, six-, and twelve-month follow-up.
  Defined as a change in a patient's depressive status from an initial score above the cutoff (PHQ-9 ≥ 10) and a follow-up score below this reference value (PHQ-9 < 10).
Health-related quality of life | Three-, six-, and twelve-month follow-up.
  Defined as a patient's score on the scales and main components of the Short-Form 12 Health Survey (SF-12).
  The SF-12 minimum and maximum values are 0 and 100 points. Higher scores mean better outcomes.
Social solving problem skills | Three-, six-, and twelve-month follow-up.
  Defined as a patient's score on the Positive Problem Orientation and Rational Problem Solving Style subscales of the Social Problem-Solving Inventory - Revised Short Form (SPSI-R:S).
  The SPSI-R:S minimum and maximum values are 0 and 100 points. Higher scores on the Positive Problem Orientation and the Rational Problem Solving Style, and lower scores on the Negative Problem Orientation, Impulsivity/Carelessness Style, and Avoidance Style mean better outcomes.
Proportion of participants with change in blood pressure | Three-, six-, and twelve-month follow-up.
  Defined as the achievement of therapeutic goal in the normalization of blood pressure according to the national standards established in the Clinical Guidelines of Primary or Essential Arterial Hypertension in people aged 15 or older. The therapeutic goal is to attain a value lower than 140/90 mmHg in non-diabetic patients and lower than 130/80 mmHg in patients with very high cardiovascular risk, diabetes, and/or proteinuric nephropathy. These values will be obtained from the patients' clinical records.
Ad-hoc questionnaire for the assessment of the acceptability of depression treatment | Three-, six-, and twelve-month follow-up.
  The ad-hoc instrument for evaluating the acceptability of the interventions is a self-report questionnaire that consists in 12 Likert-type items with four answer choices ranging from 1 (strongly agree) to 4 (strongly disagree). The construction of this instrument was based on the theoretical framework of acceptability, proposed by Sekhon et al., which characterizes seven dimensions for this concept: ethicality, affective attitude, burden, opportunity costs, perceived effectiveness, self-efficacy, and intervention coherence. For their interpretation, the participants' scores will be transformed into percentages (0% to 100%), with higher values representing more intervention acceptability.
Proportion of participants with change in glycosylated hemoglobin | Three-, six-, and twelve-month follow-up.
  Defined as the achievement of glycemic control, according to the national standards established in the Clinical Guidelines for Type II Diabetes Mellitus. Maintaining levels of glycosylated hemoglobin below 7% is regarded as a therapeutic goal in type II diabetes mellitus. These values will be obtained from the patients' clinical records.

OTHER OUTCOMES:
Utilization of health care services | Three-, six-, and twelve-month follow-up.
  The questionnaire about the utilization of health care services, adapted from the Chilean National Socioeconomic Characterization Survey, has a three-month recall period and records physician consultations or treatments, primary care and/or hospital emergencies, specialist medical treatment or mental health treatment, and hospitalizations, noting the total number of sessions (total days for hospitalizations) and the payment made for each session. The minimum number of sessions or total days for hospitalizations (and payment) are 0, there is no maximum value defined. A priori, we do not know if a higher number of sessions (consultations) mean a better or worse outcome. However, a higher humber of hospitalization days and higher payment mean worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Graciela Rojas, Principal Investigator — University of Chile
Locations (1):
- Dirección de Salud Municipal I. Municipalidad de El Bosque, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rojas G, Martinez P, Guajardo V, Campos S, Herrera P, Vohringer PA, Gomez V, Szabo W, Araya R. A collaborative, computer-assisted, psycho-educational intervention for depressed patients with chronic disease at primary care: protocol for a cluster randomized controlled trial. BMC Psychiatry. 2021 Aug 21;21(1):418. doi: 10.1186/s12888-021-03380-2. PMID 34419010